CLINICAL TRIAL: NCT05674253
Title: Combined Use of Dexmedetomidine and Hydrocortisone to Prevent New Onset Atrial Fibrillation After Coronary Artery Bypass Grafting Surgery
Brief Title: Combined Use of Dexmedetomidine and Hydrocortisone to Prevent New Onset AF After CABG Surgery
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Alaaeldin Abdelmoneem Alhadidy, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMASU R 261/2022
Record Dates: First submitted 2022-12-30; First posted 2023-01-06 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Atrial Fibrillation New Onset
Keywords: Atrial Fibrillation; Coronary artery bypass grafting; Dexmedetomidine; Hydrocortisone
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dexmedetomidine; Hydrocortisone; hydrocortisone hemisuccinate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine + Hydrocortisone group (Active Comparator): Patients will receive dexmedetomidine 0.7 ɥg/kg/hr IV infusion before aortic cross-clamping, and will be continued intra-operatively and in ICU till weaning from mechanical ventilation Patients also will also receive Hydrocortisone 100 mg intravenous (IV) before aortic cross-clamping then 100 mg every 8 hours after surgery which will be continued for 48 hours .
  Interventions: Drug: Dexmedetomidine + Hydrocortisone
- Standard group (No Intervention): Patients will not receive dexmedetomidine nor Hydrocortisone and will receive the standard management

INTERVENTIONS:
Drug: Dexmedetomidine + Hydrocortisone — Patients will receive dexmedetomidine 0.7 ɥg/kg/hr IV infusion before aortic cross-clamping, and will be continued intra-operatively and in ICU till weaning from mechanical ventilation Patients also will also receive Hydrocortisone 100 mg intravenous (IV) before aortic cross-clamping then 100 mg every 8 hours after surgery which will be continued for 48 hours
  Other Names: Medrelaxmidine + Solu-cortef
  Arms: Dexmedetomidine + Hydrocortisone group

SUMMARY:
Atrial fibrillation (AF) occurs in 20% to 40% of patients after Coronary artery bypass grafting (CABG) and is associated with numerous detrimental sequelae. In postoperative period, the patient may be exposed to several proarrhythmogenic factors as increased endogenous catecholamines, inflammatory and oxidative mediators secondary to surgical stress and the systemic response to cardiopulmonary bypass, use of inotropic support. Steroids suppress the release of the above-mentioned inflammatory mediators. Dexmedetomidine is sympatholytic, along with anti-inflammatory properties. so combined use of both drugs may have synergistic effect to prevent post operative AF (POAF)

DETAILED DESCRIPTION:
Postoperative atrial fibrillation (POAF) is a common postoperative complication that occurs in 20% to 40% of patients after Coronary artery bypass grafting (CABAG) and is associated with numerous detrimental sequelae.

POAF is an independent predictor of numerous adverse outcomes, including a 2- to 4-fold increased risk of stroke, reoperation for bleeding, infection, renal or respiratory failure, cardiac arrest, cerebral complications, need for permanent pacemaker placement, and a 2-fold increase in all-cause 30-day and 6-month mortality.

Clinical efforts to prevent and manage POAF following cardiac surgery have thus far presented a major challenge and results have been less than optimal. Despite numerous trials examining prophylactic and treatment modalities, POAF incidence following cardiac surgery has not changed over the past several decades.

The pathogenesis of POAF is incompletely understood but likely involves interplay between pre-existing physiological components and local and systemic inflammation. cardiopulmonary bypass and ischemia/reperfusion injury triggers generalized response characterized by leukocyte and complement activation, high levels of C-reactive protein (CRP) complexes, as well high levels of inflammatory mediators. These mediators, such as interleukins-6 and -8, tumor necrosis factors, leukotriene B4, and tissue plasminogen activator, might contribute to many postoperative complications including atrial fibrillation (AF).

Because of the known physiologic effects of steroids to suppress the release of the above-mentioned inflammatory mediators, steroids might have beneficial effects in decreasing postoperative AF, and inhibiting the inflammatory process post cardiopulmonary bypass. Moreover, they decrease capillary wall permeability, preventing migration of inflammatory mediators into the systemic circulation. Also, Corticosteroids decrease the heterogeneity of atrial conduction and reduce inflammation following cardiac surgery, and studies have shown that preoperative prophylactic corticosteroids reduced POAF incidence without an increased rate of postoperative infection.

Dexmedetomidine is a very specific intravenously and short-acting alpha-2 agonist which theoretically reduces the sympathetic output by decreasing serum levels of norepinephrine and inhibits the release of cytokines and results in reduction of the incidence of tachycardia, inflammation, high blood pressure during and after surgery. Dexmedetomidine reduces heart rate and consequently improves myocardial oxygen demand. It also depresses sinus node and atrial ventricular nodal function which, along with the drug's anti-inflammatory properties, makes dexmedetomidine a reasonable prophylactic drug for postoperative atrial fibrillation.

So, the investigators that combined use of both drugs will have synergistic effect to prevent (POAF) after (CABG) surgery.

ELIGIBILITY:
Inclusion Criteria:

- Scheduled for CABG Surgery with cardiopulmonary bypass (CPB) pump

Exclusion Criteria:

* History of heart block.
* Patients with preoperative bradycardia (HR < 60 / min)
* Patients with preoperative hypotension (systolic blood pressure < 90 mmhg)
* Previous episodes of AF or flutter.
* Uncontrolled diabetes mellitus requiring insulin treatment with recent hyperglycemia which required hospital treatment.
* History of peptic ulcer disease.
* Active systemic bacterial or mycotic infection.
* Permanent pacemaker.
* Any documented or suspected supraventricular or ventricular arrhythmias.
* Urgent or emergency surgery.
* Planned off-pump surgery.
* Patient Refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2022-12-25 (Actual); Primary Completion 2023-06-25 (Estimated); Study Completion 2023-07-25 (Estimated)

PRIMARY OUTCOMES:
Occurrence of AF | Up to 7 days Postoperative
  The occurrence of an episode of AF postoperatively

SECONDARY OUTCOMES:
ICU stay | Up to 7 days Postoperative
  length of ICU stay in days
Hospital stay | Up to 10 days Postoperative
  length of hospital stay in days
Bradycardia | Up to 2 days Postoperative
  Occurrence of Bradycardia defined as: HR≤50 bpm
Hypotension | Up to 2 days Postoperative
  Occurrence of Hypotension defined as decrease in systolic blood pressure >20%of basal
Hyperglycemia | Up to 7 days Postoperative
  Occurrence of Uncontrolled hyperglycemia Defined as insulin requirement >1 units/kg/day or > 100 units/day of insulin to keep RBS < 180 mg/dL
Wound infection | Up to 2 weeks Postoperative
  The occurrence of Wound infection postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiothoracic Academy, Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shen J, Lall S, Zheng V, Buckley P, Damiano RJ Jr, Schuessler RB. The persistent problem of new-onset postoperative atrial fibrillation: a single-institution experience over two decades. J Thorac Cardiovasc Surg. 2011 Feb;141(2):559-70. doi: 10.1016/j.jtcvs.2010.03.011. PMID 20434173
- [Background] Greenberg JW, Lancaster TS, Schuessler RB, Melby SJ. Postoperative atrial fibrillation following cardiac surgery: a persistent complication. Eur J Cardiothorac Surg. 2017 Oct 1;52(4):665-672. doi: 10.1093/ejcts/ezx039. PMID 28369234
- [Background] Liu C, Wang J, Yiu D, Liu K. The efficacy of glucocorticoids for the prevention of atrial fibrillation, or length of intensive care unite or hospital stay after cardiac surgery: a meta-analysis. Cardiovasc Ther. 2014 Jun;32(3):89-96. doi: 10.1111/1755-5922.12062. PMID 24495440
- [Background] Philip I, Berroeta C, Leblanc I. Perioperative challenges of atrial fibrillation. Curr Opin Anaesthesiol. 2014 Jun;27(3):344-52. doi: 10.1097/ACO.0000000000000070. PMID 24633361
- [Background] Narisawa A, Nakane M, Kano T, Momose N, Onodera Y, Akimoto R, Kobayashi T, Iwabuchi M, Okada M, Miura Y, Kawamae K. Dexmedetomidine sedation during the nighttime reduced the incidence of postoperative atrial fibrillation in cardiovascular surgery patients after tracheal extubation. J Intensive Care. 2015 May 30;3(1):26. doi: 10.1186/s40560-015-0092-5. eCollection 2015. PMID 26060574
- [Background] Keating GM. Dexmedetomidine: A Review of Its Use for Sedation in the Intensive Care Setting. Drugs. 2015 Jul;75(10):1119-30. doi: 10.1007/s40265-015-0419-5. PMID 26063213
- [Background] Ueki M, Kawasaki T, Habe K, Hamada K, Kawasaki C, Sata T. The effects of dexmedetomidine on inflammatory mediators after cardiopulmonary bypass. Anaesthesia. 2014 Jul;69(7):693-700. doi: 10.1111/anae.12636. Epub 2014 Apr 28. PMID 24773263
- [Background] January CT, Wann LS, Calkins H, Chen LY, Cigarroa JE, Cleveland JC Jr, Ellinor PT, Ezekowitz MD, Field ME, Furie KL, Heidenreich PA, Murray KT, Shea JB, Tracy CM, Yancy CW. 2019 AHA/ACC/HRS Focused Update of the 2014 AHA/ACC/HRS Guideline for the Management of Patients With Atrial Fibrillation: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2019 Jul 9;74(1):104-132. doi: 10.1016/j.jacc.2019.01.011. Epub 2019 Jan 28. No abstract available. PMID 30703431
- [Background] Leung L, Lee LHN, Lee B, Chau A, Wang EHZ. The safety of high-dose dexmedetomidine after cardiac surgery: a historical cohort study. Can J Anaesth. 2022 Mar;69(3):323-332. doi: 10.1007/s12630-021-02167-z. Epub 2021 Dec 29. PMID 34966972
- [Background] Al-Shawabkeh Z, Al-Nawaesah K, Anzeh RA, Al-Odwan H, Al-Rawashdeh WA, Altaani H. Use of short-term steroids in the prophylaxis of atrial fibrillation after cardiac surgery. J Saudi Heart Assoc. 2017 Jan;29(1):23-29. doi: 10.1016/j.jsha.2016.03.005. Epub 2016 Apr 7. PMID 28127215
- [Background] Church TJ, Haines ST. Treatment Approach to Patients With Severe Insulin Resistance. Clin Diabetes. 2016 Apr;34(2):97-104. doi: 10.2337/diaclin.34.2.97. PMID 27092020
- [Background] Engelman DT, Ben Ali W, Williams JB, Perrault LP, Reddy VS, Arora RC, Roselli EE, Khoynezhad A, Gerdisch M, Levy JH, Lobdell K, Fletcher N, Kirsch M, Nelson G, Engelman RM, Gregory AJ, Boyle EM. Guidelines for Perioperative Care in Cardiac Surgery: Enhanced Recovery After Surgery Society Recommendations. JAMA Surg. 2019 Aug 1;154(8):755-766. doi: 10.1001/jamasurg.2019.1153. PMID 31054241
- [Derived] Alhadidy MA, Alansary AM, Elghareeb SH. Combined Use of Dexmedetomidine and Hydrocortisone to Prevent New-Onset Atrial Fibrillation After Coronary Artery Bypass Grafting Surgery: A Randomized Clinical Trial. Semin Cardiothorac Vasc Anesth. 2025 Dec;29(4):284-290. doi: 10.1177/10892532251338374. Epub 2025 Apr 27. PMID 40289414